CLINICAL TRIAL: NCT07078786
Title: Comparison of Effect of Antenatal Dexamethasone Versus Betamethasone on Antepartum Cardiactocography
Brief Title: Effect of Pre-delivery Dexamethasone in Comparison With Betamethasone on Fetal Heart Trace
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rawalpindi Medical College (Other)
Collaborators: Rawalpindi Medical College, Pakistan (Other)
Responsible Party: Principal Investigator, Ifra Shafique, Principal Investigator, Rawalpindi Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1080/IREF/RMU/2024
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cardiotocography; Steroids
Keywords: Antenatal Steroids; Fetal Cardiotocography; Risk of Pre-term birth
MeSH Terms: interventions — betamethasone sodium phosphate; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomly divided into two groups using computer generated numbers and will be masked to the treatment they receive. The person assessing outcome i.e. fetal cardiotography activity will be masked to the treatment participant received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group Betamethasone (Experimental): Intramuscular injection of Betamethasone 12mg will be administered on 2 consecutive days
  Interventions: Drug: Betamethason Sodium Phosphate
- Group Dexmaethasone (Active Comparator): 24mg of Dexamethasone in two divided doses will be given Intramuscularly over 24 hours apart
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Betamethason Sodium Phosphate — Intramuscular injection of Betamethasone 12mg will be administered on 2 consecutive days
  Arms: Group Betamethasone
Drug: Dexamethasone — two doses of 12mg of IM Dexamethasone given 24 hours apart
  Arms: Group Dexmaethasone

SUMMARY:
As baby grows inside the womb of mother, heart and other organs develop. The heart activity can be recorded by placing a transducer on the belly of mother. The tracing obtain provides information about heart rate, any increase or decrease in heart rate and how much it varies with time. Variation in heart rate along with increase is indicator of fetal well being. Some mothers are at high risk of pre-term birth that is baby delivery before 37 weeks of gestation. In such cases steroids are given to mother to accelerate lung development of the baby so that it can easily adapt to outside world. Dexamethasone and Betamethasone are commonly used steroids which can also effect fetal heart activity.

DETAILED DESCRIPTION:
Some patients are at high risk of Pre term birth and therefore they are advised antenatal steroids which facilitates fetal lung development preparing it for smoother transition for extra-uterine life. Dexamethasone and Betamethasone are commonly used for this purpose but differently effect fetal cardiac activity as evident by CTG changes and awareness of these phenomena would prevent iatrogenic delivery of preterm fetuses.

ELIGIBILITY:
Inclusion Criteria:

* History of pre term labor
* Preterm pre labor rupture of membranes
* Third trimester bleeding due to placenta previa

Exclusion Criteria:

* IUGR
* Uteroplacental insufficiency
* Oligohydroamnios
* Maternal drug therapy that can effect fetal heart rate
* Contraindications to Intramuscular injections
* Patients admitted with non reassuring CTG

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant Females with Gestational age 30-37 weeks are included in the study
Enrollment: 110 (Estimated)
Dates: Start 2025-07-13 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Mean number of accelerations on fetal cardiotocography | Before intervention, 2 and 4 days after intervention
Long term heart rate variability on fetal cardiotocography | Before intervention, 2 and 4 days after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ifra Shafique, MBBS, Principal Investigator — Rawalpindi Medical Unviersity
Locations (1):
- Holy Family Hospital, Rawalpindi Medical University, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rotmensch S, Liberati M, Vishne TH, Celentano C, Ben-Rafael Z, Bellati U. The effect of betamethasone and dexamethasone on fetal heart rate patterns and biophysical activities. A prospective randomized trial. Acta Obstet Gynecol Scand. 1999 Jul;78(6):493-500. PMID 10376858
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/10376858/